CLINICAL TRIAL: NCT05838274
Title: Biological Risk Factors for the Prospective Development of Alcohol Use Disorders in Young Adults With Bipolar Disorder and Typically Developing Young Adults
Brief Title: Acute Alcohol Response In Bipolar Disorder: a Longitudinal Alcohol Administration/fMRI Study
Acronym: Long_BACS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Elizabeth Thomas Cox Lippard, Associate Professor, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: R01AA030038 (NIH)
Record Dates: First submitted 2023-04-10; First posted 2023-05-01 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Bipolar Disorder; Alcohol Drinking; Alcohol Use Disorder
MeSH Terms: conditions — Bipolar Disorder; Alcohol Drinking; Alcoholism | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol (Active Comparator): Participants will be provided alcohol during study visits and changes in behavior/neural activity after consuming alcohol will be examined.
  Interventions: Other: Alcohol vs. Placebo beverage conditions
- Placebo (Placebo Comparator): placebo beverage condition
  Interventions: Other: Alcohol vs. Placebo beverage conditions

INTERVENTIONS:
Other: Alcohol vs. Placebo beverage conditions — Individuals will drink beverages containing alcohol. How they respond to a high vs. low dose will be compared.

SUMMARY:
Alcohol use disorders (AUDs) affect up to 60% of individuals with bipolar disorder during their lifetime and is associated with worse illness outcomes, yet few studies have been performed to clarify the causes of this comorbidity. Understanding biological risk factors that associate with and predict the development of AUDs in bipolar disorder could inform interventions and prevention efforts to reduce the rate of this comorbidity and improve outcomes of both disorders. Identifying predictors of risk requires longitudinal studies in bipolar disorder aimed at capturing the mechanisms leading to the emergence of AUDs. Previous work in AUDs suggest that subjective responses to alcohol and stress-related mechanisms may contribute to the development of AUDs. In bipolar disorder, altered developmental trajectory of critical ventral prefrontal networks that modulate mood and reward processing may alter responses to alcohol and stressors; consequently, the disruption in typical neurodevelopment may be an underlying factor for the high rates of comorbidity. No longitudinal data exist investigating if this developmental hypothesis is correct. To address this gap, the investigators will use a multimodal neuroimaging approach, modeling structural and functional neural trajectories of corticolimbic networks over young adulthood, incorporating alcohol administration procedures, clinical phenotyping, and investigating effects of acute stress exposure and early life stress. Research aims are to identify biological risk factors-i.e., changes in subjective response to alcohol and associated neural trajectories-that are associated with the development of alcohol misuse and symptoms of AUDs over a two-year longitudinal period in young adults with bipolar disorder and typical developing young adults. Longitudinal data will be collected on 160 young adults (50% with bipolar disorder, 50% female; aged 21-26). This study is a natural extension of the PI's K01 award. How acute exposure to stress and childhood maltreatment affects subjective response to alcohol and risk for prospective alcohol misuse and symptoms of AUDs will be investigated. The investigators will test our hypothesis that developmental differences in bipolar disorder versus typical developing individuals disrupt corticolimbic networks during young adulthood, increase sensitivity to stress, and lead to changes in subjective response to alcohol and placebo response increasing risk for developing AUDs.

DETAILED DESCRIPTION:
The PI is currently investigating subjective response to alcohol in bipolar disorder and typical developing young adults (n=60; 50% with bipolar disorder) using placebo-controlled alcohol administration with baseline structural/functional MRI assessments collected with her K01. The proposed work will extend this active study to enroll 100 new young adults (50% with bipolar disorder) to complete baseline clinical, MRI, and placebo-controlled alcohol administration sessions. The PI's K01 is focused on investigating differences in subjective and neural response to alcohol between bipolar disorder and typical developing young adults. The proposed study will focus on investigating changes in subjective response to alcohol, placebo response, and relations with neural trajectories, the role(s) of stress, and prediction of alcohol problems over a two-year period. Longitudinal follow-up (clinical, detailed assessment of alcohol use, and MRI) will occur on average 1- and 2-years following enrollment. Participants enrolled on the PI's K01 will be brought back for longitudinal assessments to reach N=80 per group with longitudinal data (50% female; aged 21-26)]. At 2-year follow-up, placebo-controlled alcohol administration sessions will be repeated to test if sensitivity to alcohol changes over time-and if change in sensitivity to alcohol is associated with progressive neural changes in corticolimbic brain networks during young adulthood-and associations with alcohol use and symptoms of AUDs over time, and interactions with bipolar disorder. Changes in placebo-response and if changes are predictive of increased alcohol use and symptoms of AUDs will also be modeled. At one-year follow-up, a subset of participants will be invited to complete a psychosocial stress and neutral fMRI task on separate days (counter balanced; n=40 per group). Participants will immediately complete an alcohol session following the fMRI tasks and stress-induced changes in subjective response to alcohol and interactions with group will be modeled.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for all participants:

* between 21 and 26 years of age
* having consumed at least 4 (men) or 3 (women) drinks on a single occasion over the last year
* euthymic at the time of enrollment

Inclusion criteria for bipolar disorder participants:

- Meeting Diagnostic and Statistical Manual-5 Research Version (DSM-V-RV) diagnostic criteria for bipolar disorder, confirmed by structured interview

Exclusion Criteria:

For all subjects exclusion criteria include:

* history of significant medical illness, particularly if possible changes in cerebral tissue
* neurologic abnormality including significant head trauma (loss of consciousness of ≥5-min)
* full Scale intelligence quotient (IQ) <85
* contraindication to MRI scanning
* positive pregnancy test
* current cannabis use disorder>moderate
* history of severe AUDs
* scores > 15 on the alcohol Use Disorders Identification Test (AUDIT; part of phone screen)
* ever being in an abstinence-oriented treatment program for alcohol use
* reporting wanting to quit drinking but not being able to
* any medical, religious, or other reasons for not drinking alcohol
* history of heart attack, heart trouble, high blood pressure, diabetes, or liver disease
* an adverse reaction to alcoholic beverages
* reporting never consuming 4 (men) or 3 (women) or more drinks on a single occasion over the last year
* unwillingness to have a friend or family member drive them home after the alcohol administration sessions
* a past year substance use disorder (other than alcohol, cannabis, or nicotine)

Additional exclusion criteria for bipolar disorder participants:

- not taking medications for greater than or equal to 4 weeks (i.e. participants must be stable on medications)

Additional exclusion criteria for healthy comparison subjects also include:

* any prior psychiatric hospitalizations
* lifetime history of a neurodevelopmental disorder, affective disorder, psychotic disorder, eating disorder
* greater than 1 month of lifetime psychotropic medication.

Ages: 21 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
changes in subjective response | 2 years
  Subjective response to alcohol will be measured with the subjective effects of alcohol scale (SEAS) at baseline and two-years later and changes in subjective response to alcohol over time (SEAS two year follow-up minus SEAS baseline) investigated and interactions with group (young adults with bipolar disorder, typical comparison young adults) modeled.
Neural trajectories associated with subjective response to alcohol | 2 years
  Changes in neural trajectories over the two-year follow-up period will be modeled and relations with subjective response at two-year follow-up investigated. We will model changes in cortical thickness and surface area of frontolimbic regions of interest and investigate if these neural trajectories relate to changes in subjective response to alcohol (measured with the SEAS at baseline and follow-up).
Relations between changes in subjective response and associated neural trajectories with alcohol use disorder symptoms at two-year follow-up | 2 years
  Changes in subjective response (measured with the SEAS) and neural trajectories over the follow up period (changes in cortical thickness and surface area of frontlimbic regions of interest) and relations with alcohol problems at two-year follow up will be modeled with number of alcohol use disorder symptoms on the SCID at two-year follow up as the dependent variable.
Relations between changes in subjective response and associated neural trajectories with alcohol misuse and problems at two-year follow-up | 2 years
  Changes in subjective response (measured with the SEAS) and neural trajectories over the follow up period (changes in cortical thickness and surface area of frontolimbic regions of interest) and relations with alcohol problems at two-year follow up will be modeled with AUDIT score at two-year follow up as the dependent variable.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Lippard, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
After study completion and publication of finding, functional neuroimaging data and behavior data collected following alcohol and placebo conditions will be shared.
Supporting Information: SAP
Time Frame: We will complete all our analyses and publish results and methodologies in scientific journals before the data are available to the research community. Data will be made available following 6 months after publication.
Access Criteria: We will be collecting identifying information. Even though the final dataset will be stripped of identifiers prior to release for sharing, we believe that there remains the possibility of deductive disclosure of subjects with unusual characteristics. Thus, we will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.